CLINICAL TRIAL: NCT07289230
Title: A Comparative Study Between Sheathless RIRS, Traditional Access Sheath RIRS, and Suction Access Sheath RIRS in the Management of Renal Stones ≤ 2 cm: A Randomized Controlled Clinical Trial
Brief Title: Sheathless, Traditional, and Suction Access Sheath RIRS for Renal Stones ≤2 cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, AbdAlhameed Naser, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU_MS400_2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Kidney Calculi; Renal Calculi; Urolithiasis; Nephrolithiasis
Keywords: Kidney stones; Renal calculi; Urolithiasis; Endoscopic management of kidney stones; Retrograde intrarenal surgery; Flexible ureterorenoscopy; Ureteral access sheath; Suction ureteral access sheath; Sheathless retrograde intrarenal surgery; Minimally invasive urologic surgery
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a parallel fashion to one of three study arms: traditional ureteral access sheath retrograde intrarenal surgery (RIRS), suction ureteral access sheath retrograde intrarenal surgery (RIRS), or sheathless retrograde intrarenal surgery (RIRS). Each participant received only one of the three techniques, and the groups were followed and compared concurrently regarding stone clearance, operative time, intraoperative complications, and early postoperative complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Ureteral Access Sheath Retrograde Intrarenal Surgery (Active Comparator): Participants in this arm underwent retrograde intrarenal surgery (retrograde intrarenal surgery) using a traditional ureteral access sheath. A flexible ureteroscope was advanced through an 11 French by 13 French ureteral access sheath positioned near the ureteropelvic junction. Irrigation was maintained at 50 to 100 milliliters per minute. Stone fragmentation was performed using a holmium:yttrium-aluminum-garnet laser device. All patients received a six French double-J stent at the end of the procedure. Intraoperative complications were recorded, and postoperative imaging was performed for outcome assessment.
  Interventions: Procedure: Traditional ureteral access sheath retrograde intrarenal surgery
- Suction Ureteral Access Sheath Retrograde Intrarenal Surgery (Experimental): Participants in this arm underwent retrograde intrarenal surgery (retrograde intrarenal surgery) with the use of a suction ureteral access sheath. An 11 French suction ureteral access sheath was inserted over a guidewire and positioned in the renal pelvis. The suction system was connected to a vacuum device, with negative pressure set between 2 and 7 kilopascals to facilitate evacuation of stone fragments and reduce intrarenal pressure. The same flexible ureteroscope and holmium:yttrium-aluminum-garnet laser lithotripsy technique were used as in the traditional arm. A six French double-J stent was inserted at the end of the operation. All intraoperative and postoperative findings were documented.
  Interventions: Procedure: Suction ureteral access sheath retrograde intrarenal surgery
- Sheathless Retrograde Intrarenal Surgery (Experimental): Participants in this arm underwent sheathless retrograde intrarenal surgery (retrograde intrarenal surgery), in which the flexible ureteroscope was inserted directly over a guidewire without the placement of any ureteral access sheath. Stone fragmentation was performed using a holmium:yttrium-aluminum-garnet laser device. A six French double-J stent was placed at the end of the procedure. Any intraoperative complications, such as bleeding or extravasation, were documented, and postoperative imaging was conducted to assess stone clearance.
  Interventions: Procedure: Sheathless retrograde intrarenal surgery

INTERVENTIONS:
Procedure: Traditional ureteral access sheath retrograde intrarenal surgery — This intervention involves performing retrograde intrarenal surgery using a traditional ureteral access sheath to facilitate entry of the flexible ureteroscope and maintain controlled intrarenal pressure. The procedure includes endoscopic fragmentation of renal calculi using a holmium:yttrium-aluminum-garnet laser device and placement of a double-J ureteral stent at the end of surgery.
  Arms: Traditional Ureteral Access Sheath Retrograde Intrarenal Surgery
Procedure: Suction ureteral access sheath retrograde intrarenal surgery — This intervention uses a suction ureteral access sheath that provides continuous negative pressure during retrograde intrarenal surgery. The system assists in evacuation of stone debris and helps control intrarenal pressure while the flexible ureteroscope and holmium:yttrium-aluminum-garnet laser device are used for stone fragmentation. A double-J ureteral stent is placed after the procedure.
  Arms: Suction Ureteral Access Sheath Retrograde Intrarenal Surgery
Procedure: Sheathless retrograde intrarenal surgery — This intervention involves performing retrograde intrarenal surgery without the use of any ureteral access sheath. The flexible ureteroscope is introduced directly over a guidewire to access the renal collecting system for laser fragmentation of the stone using a holmium:yttrium-aluminum-garnet laser device. A double-J ureteral stent is inserted following completion of the procedure.
  Arms: Sheathless Retrograde Intrarenal Surgery

SUMMARY:
This completed randomized clinical study was designed to compare three different techniques of retrograde intrarenal surgery (retrograde intrarenal surgery) for the treatment of kidney stones that are 2 centimeters or smaller. Retrograde intrarenal surgery is a minimally invasive procedure in which a flexible scope is passed through the urinary tract to reach the kidney and fragment the stone.

The clinical study included three groups of patients. The first group underwent retrograde intrarenal surgery using a traditional ureteral access sheath, which is a hollow tube placed in the ureter to facilitate the passage of instruments and help control pressure inside the kidney. The second group underwent retrograde intrarenal surgery using a suction ureteral access sheath, which combines the function of a traditional sheath with gentle suction to help remove stone fragments and reduce internal pressure. The third group underwent sheathless retrograde intrarenal surgery, in which the flexible surgical scope is inserted directly without the use of any ureteral access sheath.

The purpose of this clinical study was to determine whether these three approaches differ in terms of stone clearance, operative time, intraoperative complications such as bleeding or fluid leakage, and early postoperative complications such as fever or infection. All participants were adults with a single kidney stone between 1 and 2 centimeters, normal kidney function, and no active infection or anatomical abnormalities. All procedures were performed at Ain Shams University Hospitals using the same surgical equipment and technique to ensure comparability between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Symptomatic unilateral single renal stone with a maximal diameter from 1 centimeter to 2 centimeters.
* Normal kidney function based on routine laboratory tests.
* Patients willing and able to provide written informed consent to participate in the clinical study.

Exclusion Criteria:

* Patients with active urinary tract infection (UTI) until appropriate treatment is completed and infection is cleared.
* Patients with anatomical abnormalities of the urinary tract (for example, congenital or acquired structural abnormalities).
* Pregnant patients.
* Patients who are medically unfit for general anesthesia.
* Patients with multiple renal stones in the same kidney or bilateral renal stones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Stone-free rate assessed by non-contrast computed tomography of the urinary tract | One month after surgery (non-contrast computed tomography of the urinary tract performed approximately 30 days postoperatively)
  Stone-free status is evaluated using non-contrast computed tomography of the urinary tract performed after surgery. Residual stone fragments are classified into four grades: Grade A, no stones detected (absolute stone-free); Grade B, residual fragments less than or equal to 2 millimeters (relative stone-free); Grade C, residual fragments 2.1 to 4 millimeters (relative stone-free); and Grade D, residual fragments greater than 4 millimeters (significant residual stones). The primary endpoint is the proportion of patients achieving stone-free status, defined as Grade A (absolute stone-free) and, in a secondary analysis, Grades A to C combined (clinically insignificant residual fragments).

SECONDARY OUTCOMES:
Operative time for retrograde intrarenal surgery | During the surgical procedure on the day of surgery
  Operative time is measured in minutes from the insertion of the endoscopic instruments at the beginning of retrograde intrarenal surgery until completion of the procedure, including placement of the double-J ureteral stent. The metric is the mean operative time and distribution of operative time for each study arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals - Department of Urology, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results of the completed clinical study will be made available to qualified researchers upon reasonable request. Shared data will include de-identified clinical information related to baseline characteristics, operative details, postoperative outcomes, and imaging-based assessments. No information that could directly identify a participant will be shared. Data will be provided for the purpose of scientific validation, secondary analysis, or meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data and supporting documents will become available beginning six months after publication of the study results and will remain available for a period of five years following that date.
Access Criteria: Researchers wishing to access the de-identified dataset must submit a written request outlining their study objectives and analysis plan. Requests will be evaluated by the study investigators to ensure scientific validity and appropriate use of the data. Approved researchers will be required to sign a data use agreement stating that the information will be used solely for research purposes, will not be shared with unauthorized parties, and will not be used in any attempt to identify study participants.